CLINICAL TRIAL: NCT02951026
Title: A Phase 3, Multicenter, Observational Long-term Study Evaluating the Safety, Tolerability, and Efficacy of Treatment of SM04690 or Placebo Previously Injected in the Target Knee Joint of Subjects With Moderately to Severely Symptomatic Osteoarthritis
Brief Title: An Observational Study Evaluating the Safety, Tolerability, and Efficacy of Treatment of SM04690 or Placebo Previously Injected in the Target Knee Joint of Subjects With Moderately to Severely Symptomatic Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SM04690-OA-05
Record Dates: First submitted 2016-10-07; First posted 2016-11-01 (Estimated); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Osteoarthritis
Keywords: knee; osteoarthritis; intra-articular injection; SM04690
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 0.03mg SM04690 (previously injected): Subjects in this group received a single intra-articular injection of 0.03mg SM04690 into the target knee during the "parent" study prior to enrolling in this observational study.
  Interventions: Other: Not applicable (no therapy is administered as part of this study)
- 0.07mg SM04690 (previously injected): Subjects in this group received a single intra-articular injection of 0.07mg SM04690 into the target knee during the "parent" study prior to enrolling in this observational study.
  Interventions: Other: Not applicable (no therapy is administered as part of this study)
- 0.23mg SM04690 (previously injected): Subjects in this group received a single intra-articular injection of 0.23mg SM04690 into the target knee during the "parent" study prior to enrolling in this observational study.
  Interventions: Other: Not applicable (no therapy is administered as part of this study)
- Placebo (previously injected): Subjects in this group received a single intra-articular injection of placebo into the target knee during the "parent" study prior to enrolling in this observational study.
  Interventions: Other: Not applicable (no therapy is administered as part of this study)

INTERVENTIONS:
Other: Not applicable (no therapy is administered as part of this study) — No experimental therapy or placebo is being administered in this study. All subjects in this observational study received a single intra-articular injection of SM04690 or placebo in a prior "parent" study.

SUMMARY:
This long-term extension study is designed to monitor the long-term safety, tolerability, and efficacy of treatment of SM04690 or placebo previously injected in the target knee joints of subjects with moderately to severely symptomatic osteoarthritis (OA) from a Samumed-sponsored SM04690-OA phase 2 or phase 3 study. No additional SM04690 or placebo therapy will be administered in this study.

ELIGIBILITY:
Inclusion Criteria:

* Completion of scheduled end-of-study visit of Samumed-sponsored SM04690-OA phase 2 or phase 3 studies
* Full understanding of the requirements of the study and willingness to comply with all study visits and assessments
* Subjects must have read and understood the informed consent form, and must have signed it prior to any study-related procedure being performed

Exclusion Criteria:

* Unable to undergo the radiograph procedures detailed within the protocol
* Partial or complete joint replacement in the target knee
* Subjects who are immediate family members (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study at the investigative site, or are directly affiliated with the study at the investigative site
* Subjects employed by Samumed, LLC, or any of its affiliates or development partners (that is, an employee, temporary contract worker, or designee) responsible for the conduct of the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects can only participate in this study upon completion of a Samumed SM04690-OA phase 2 or phase 3 study.
Sampling Method: Probability Sample
Enrollment: 703 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence rate of serious adverse events (SAEs) | Month 60
  Compare the incidence rate of SAEs occurring in the (previously injected) SM04690 treatment arms to the (previously injected) placebo treatment arm by Month 60

SECONDARY OUTCOMES:
Adverse events (AEs) of interest | Month 6
  Compare the number of subjects who experience an AE of interest occurring in the (previously injected) SM04690 treatment arms to the (previously injected) placebo treatment arm at Month 6. AEs of interest include those related to either knee and/or an AE that is a newly diagnosed chronic condition requiring treatment (e.g., hypertension, hyperlipidemia, diabetes).
AEs of interest | Month 12
  Compare the number of subjects who experience an AE of interest occurring in the (previously injected) SM04690 treatment arms to the (previously injected) placebo treatment arm at Month 12.
AEs of interest | Month 24
  Compare the number of subjects who experience an AE of interest occurring in the (previously injected) SM04690 treatment arms to the (previously injected) placebo treatment arm at Month 24.
AEs of interest | Month 36
  Compare the number of subjects who experience an AE of interest occurring in the (previously injected) SM04690 treatment arms to the (previously injected) placebo treatment arm at Month 36.
AEs of interest | Month 48
  Compare the number of subjects who experience an AE of interest occurring in the (previously injected) SM04690 treatment arms to the (previously injected) placebo treatment arm at Month 48.
AEs of interest | Month 60
  Compare the number of subjects who experience an AE of interest occurring in the (previously injected) SM04690 treatment arms to the (previously injected) placebo treatment arm at Month 60.
Incidence and incidence rate of total knee replacement (TKR) | Month 60
  Compare the incidence and incidence rate of TKR in the previously injected knee occurring in the (previously injected) SM04690 treatment arms to the (previously injected) placebo treatment arm by Month 60.
Change in joint space width (JSW) | Baseline and Month 6
  Change from baseline in JSW as documented by X-ray of the target knee in both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 6.
Change in joint space width (JSW) | Baseline and Month 12
  Change from baseline in JSW as documented by X-ray of the target knee in both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 12.
Change in joint space width (JSW) | Baseline and Month 24
  Change from baseline in JSW as documented by X-ray of the target knee in both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 24.
Change in joint space width (JSW) | Baseline and Month 36
  Change from baseline in JSW as documented by X-ray of the target knee in both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 36.
Change in joint space width (JSW) | Baseline and Month 48
  Change from baseline in JSW as documented by X-ray of the target knee in both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 48.
Change in joint space width (JSW) | Baseline and Month 60
  Change from baseline in JSW as documented by X-ray of the target knee in both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 60.
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score | Baseline and Month 6
  Change from baseline in WOMAC total score for the target knee for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 6.
Change in WOMAC total score | Baseline and Month 12
  Change from baseline in WOMAC total score for the target knee for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 12.
Change in WOMAC total score | Baseline and Month 24
  Change from baseline in WOMAC total score for the target knee for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 24.
Change in WOMAC total score | Baseline and Month 36
  Change from baseline in WOMAC total score for the target knee for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 36.
Change in WOMAC total score | Baseline and Month 48
  Change from baseline in WOMAC total score for the target knee for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 48.
Change in WOMAC total score | Baseline and Month 60
  Change from baseline in WOMAC total score for the target knee for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 60.
Change in WOMAC pain subscore | Baseline and Month 6
  Change from baseline in WOMAC pain subscore for the target knee for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 6.
Change in WOMAC pain subscore | Baseline and Month 12
  Change from baseline in WOMAC pain subscore for the target knee for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 12.
Change in WOMAC pain subscore | Baseline and Month 24
  Change from baseline in WOMAC pain subscore for the target knee for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 24.
Change in WOMAC pain subscore | Baseline and Month 36
  Change from baseline in WOMAC pain subscore for the target knee for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 36.
Change in WOMAC pain subscore | Baseline and Month 48
  Change from baseline in WOMAC pain subscore for the target knee for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 48.
Change in WOMAC pain subscore | Baseline and Month 60
  Change from baseline in WOMAC pain subscore for the target knee for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 60.
Change in WOMAC function subscore | Baseline and Month 6
  Change from baseline in WOMAC function subscore for the target knee for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 6.
Change in WOMAC function subscore | Baseline and Month 12
  Change from baseline in WOMAC function subscore for the target knee for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 12.
Change in WOMAC function subscore | Baseline and Month 24
  Change from baseline in WOMAC function subscore for the target knee for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 24.
Change in WOMAC function subscore | Baseline and Month 36
  Change from baseline in WOMAC function subscore for the target knee for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 36.
Change in WOMAC function subscore | Baseline and Month 48
  Change from baseline in WOMAC function subscore for the target knee for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 48.
Change in WOMAC function subscore | Baseline and Month 60
  Change from baseline in WOMAC function subscore for the target knee for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 60.
Change in Physician Global Assessment | Baseline and Month 6
  Change from baseline OA disease activity as assessed by Physician Global Assessment for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 6.
Change in Physician Global Assessment | Baseline and Month 12
  Change from baseline OA disease activity as assessed by Physician Global Assessment for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 12.
Change in Physician Global Assessment | Baseline and Month 24
  Change from baseline OA disease activity as assessed by Physician Global Assessment for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 24.
Change in Physician Global Assessment | Baseline and Month 36
  Change from baseline OA disease activity as assessed by Physician Global Assessment for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 36.
Change in Physician Global Assessment | Baseline and Month 48
  Change from baseline OA disease activity as assessed by Physician Global Assessment for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 48.
Change in Physician Global Assessment | Baseline and Month 60
  Change from baseline OA disease activity as assessed by Physician Global Assessment for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 60.
Change in Patient Global Assessment | Baseline and Month 6
  Change from baseline OA disease activity as assessed by Patient Global Assessment for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 6.
Change in Patient Global Assessment | Baseline and Month 12
  Change from baseline OA disease activity as assessed by Patient Global Assessment for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 12.
Change in Patient Global Assessment | Baseline and Month 24
  Change from baseline OA disease activity as assessed by Patient Global Assessment for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 24.
Change in Patient Global Assessment | Baseline and Month 36
  Change from baseline OA disease activity as assessed by Patient Global Assessment for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 36.
Change in Patient Global Assessment | Baseline and Month 48
  Change from baseline OA disease activity as assessed by Patient Global Assessment for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 48.
Change in Patient Global Assessment | Baseline and Month 60
  Change from baseline OA disease activity as assessed by Patient Global Assessment for both the (previously injected) SM04690 treatment arms and the (previously injected) placebo treatment arm at Month 60.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Yazici, M.D., Study Director — Biosplice Therapeutics, Inc.
Locations (62):
- United States (62):
  - Research Site, Birmingham, Alabama
  - Research Site, Oro Valley, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Canoga Park, California
  - Research Site, Carmichael, California
  - Research Site, Cerritos, California
  - Research Site, El Cajon, California
  - Research Site, Gold River, California
  - Research Site, La Mesa, California
  - Research Site, Palm Springs, California
  - Research Site, Rancho Mirage, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Marcos, California
  - Research Site, Spring Valley, California
  - Research Site, Boulder, Colorado
  - Research Site, Stamford, Connecticut
  - Research Site, Trumbull, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, DeLand, Florida
  - Research Site, Edgewater, Florida
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Miami, Florida
  - Research Site, Marietta, Georgia
  - Research Site, Woodstock, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Newton, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Frederick, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Troy, Michigan
  - Research Site, City of Saint Peters, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Albuquerque, New Mexico
  - Research Site, Orchard Park, New York
  - Research Site, Rochester, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Knoxville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Bedford, Texas
  - Research Site, Houston, Texas
  - Research Site, San Angelo, Texas
  - Research Site, Layton, Utah
  - Research Site, Arlington, Virginia
  - Research Site, Charlottesville, Virginia

REFERENCES:
- [Derived] Swearingen CJ, Tambiah JRS, Simsek I, Ghandehari H, Kennedy S, Yazici Y. Evaluation of Safety and Efficacy of a Single Lorecivivint Injection in Patients with Knee Osteoarthritis: A Multicenter, Observational Extension Trial. Rheumatol Ther. 2025 Feb;12(1):157-171. doi: 10.1007/s40744-024-00731-9. Epub 2025 Jan 4. PMID 39755925